CLINICAL TRIAL: NCT06083259
Title: Does Cyanoacrylate Require Supportive Suturing to Reduce Seconder Bleeding and Stabilizing Biomaterial at the Donor Site?
Brief Title: Cyanoacrylate With or Without Suture?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gencay Keceli, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Palatal Wound Healing
Record Dates: First submitted 2023-09-21; First posted 2023-10-13 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Wound Heal
MeSH Terms: interventions — Sutures; Cyanoacrylates

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- gelatin sponge + cyanoacrylate + suspending sutures (Active Comparator): After administration of local anesthesia (2% articaine hydrochloride with epinephrine 1:100,000), palatal thickness will be measured by perpendicularly inserting a Michigan-O periodontal probe from the corners of the rectangular donor area. Epithelialized gingival graft will be harvested. After a rectangular-shaped initial incision, a graft with 1-1.5 mm thickness will be harvested approximately 1.5 to 3 mm away from the gingival margins of the upper teeth. The donor site will be closed with a gelatin sponge + cyanoacrylate + suspending sutures.
  Interventions: Device: Gelatin sponge stabilization with suture and cyanoacrylate
- gelatin sponge + cyanoacrylate (Active Comparator): After local anesthesia (2% articaine hydrochloride with epinephrine 1:100,000) administration, palatal thickness will be measured by perpendicularly inserting a Michigan-O periodontal probe from the corners of the rectangular donor area and the mean value will be recorded as palatal tissue thickness. The epithelialized gingival graft will be harvested using 15 knives. After a rectangular-shaped initial incision, a graft with 1-1.5 mm thickness will be harvested approximately 1.5 to 3 mm away from the gingival margins of the upper teeth. The donor site will be closed with a gelatin sponge and cyanoacrylate without sutures.
  Interventions: Procedure: Gelatin sponge stabilization with cyanoacrylate

INTERVENTIONS:
Device: Gelatin sponge stabilization with suture and cyanoacrylate — The donor site will be closed both with gelatin sponge +Cyanoacrylate (Spongostan®, Ethicon, USA)+ supporting sutures (control group)
  Arms: gelatin sponge + cyanoacrylate + suspending sutures
Procedure: Gelatin sponge stabilization with cyanoacrylate — Seconder The donor site will be closed both with gelatin sponge +Cyanoacrylate (Spongostan®, USA) (test group)
  Arms: gelatin sponge + cyanoacrylate

SUMMARY:
An epithelialized gingival graft will be harvested from the palate for the treatment of various mucogingival deformities. The donor site will be treated with either a combination of a collagen sponge and cyanoacrylate or a collagen sponge, cyanoacrylate, and suspending sutures. Intraoperatively, measurements will be taken for palatal tissue thickness, graft dimensions, working time, and primary bleeding time. Data regarding pain perception will be gauged using a visual analog scale, and the number of analgesics, secondary bleeding, epithelization level, and color match will be assessed prospectively. These outcomes will be evaluated on the first 7 days and subsequently on the 14th, 21st, and 28th days. Patient-reported outcomes will be recorded using the Oral Health Impact Profile-14 questionnaire.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

* age ≥18;
* mucogingival surgical treatment indication that needs connective tissue graft in the anterior mandible;
* stable periodontium after phase I therapy;
* full-mouth plaque and bleeding scores <15%

Exclusion Criteria:

* previous palatal harvesting history;
* unstable endodontic conditions;
* tooth mobility at the surgical site;
* systemic disease;
* pregnancy;
* use of medications with potential adverse effects on periodontal tissues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Donor site pain perception | everyday in first week
  Patients score their daily donor site pain perception using visual analog score level by giving numbers from 0 to 10 according to the visual analog scale (0: no pain, 1: minimal pain, 10: severe pain)
Secondary bleeding time | during first week
  Patients will record presence or absence of secondary bleeding (presence=1 or absence=0).

SECONDARY OUTCOMES:
Graft height | during surgery
  Dimensions will be measured during surgery by clinician using Michigan O probe (will be reported in mm)
Graft width | during surgery
  Dimensions will be measured during surgery by clinician using Michigan O probe.(will be reported in mm)
Graft thickness | during surgery
  Dimensions will be measured during surgery by clinician using Michigan O probe (will be reported in mm)
Working time | during surgery
  Harvesting process will be recorded by an blinded research assistant
Quantity of analgesics | first week
  Patients recorded the quantity of analgesics taken will be reported as quantity of pill
Sensation loss | first week, second week , third week, fourth week.
  Sensation loss will be scored by the help of clinician comparing with the symmetrical side an will be recorded as no-loss, medium loss or severe loss
Color match | first week, second week, third week, fourth week.
  Color match with the adjacent tissue was determined by researcher using a Visual Analog Pain Scale scale (0: absence of harmony, 10: excellent harmony)
Epithelization level | first week, second week, third week, fourth week.
  Epithelization level was scored by researcher as none, partial or full epithelization by means of bubble formation after dripping hydrogen peroxide (3%) to the wound surface.
The Oral Health Impact Profile-14 is a questionnaire that measures how oral disorders impact a patient's quality of life. | first week
  The questionnaire has 14 items with answers rated on a 5-point Likert scale (from 1 = never to 5 = very often) to indicate a level of different problems related to oral health

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No